CLINICAL TRIAL: NCT00072774
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of Three Fixed Doses (100 Mg, 200 Mg, Or 400 Mg) Of DVS-233 SR In Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating DVS-233 SR In Adult Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A1-306
Record Dates: First submitted 2003-11-10; First posted 2003-11-13 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Major Depressive Disorder
Keywords: Depressive Disorder, Major; Melancholia, Involutional; Depression, Involutional
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: DVS-233 SR

SUMMARY:
To compare the antidepressant efficacy and safety of subjects receiving DVS-233 SR versus subjects receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Sexually active women participating in the study must use a medically acceptable form of contraception
* Subjects must have a primary diagnosis of major depressive disorder

Exclusion Criteria:

* Treatment with DVS-233 SR at any time in the past
* Treatment with venlafaxine (immediate release [IR] or extended release [ER]) within 90 days of study day 1
* Known hypersensitivity to venlafaxine (IR or ER)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Zilcha-Mano S, Wang X, Wajsbrot DB, Boucher M, Fine SA, Rutherford BR. Trajectories of Function and Symptom Change in Desvenlafaxine Clinical Trials: Toward Personalized Treatment for Depression. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):579-584. doi: 10.1097/JCP.0000000000001435. PMID 34183490
- [Derived] Soares CN, Zhang M, Boucher M. Categorical improvement in functional impairment in depressed patients treated with desvenlafaxine. CNS Spectr. 2019 Jun;24(3):322-332. doi: 10.1017/S1092852917000633. Epub 2017 Nov 15. PMID 29140227
- [Derived] McIntyre RS, Fayyad R, Mackell JA, Boucher M. Effect of metabolic syndrome and thyroid hormone on efficacy of desvenlafaxine 50 and 100 mg/d in major depressive disorder. Curr Med Res Opin. 2016;32(3):587-99. doi: 10.1185/03007995.2015.1136603. Epub 2016 Jan 13. PMID 26709542
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. A Post Hoc Analysis of the Effect of Weight on Efficacy in Depressed Patients Treated With Desvenlafaxine 50 mg/d and 100 mg/d. Prim Care Companion CNS Disord. 2015 Jun 4;17(3):10.4088/PCC.14m01741. doi: 10.4088/PCC.14m01741. eCollection 2015. PMID 26644956
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058